CLINICAL TRIAL: NCT06558591
Title: Feasibility and Potential Impact of an Individualized Exercise Program Via a Telerehabilitation Device in Chronic Patients: A Pilot Study
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Limoges University (Other)
Collaborators: Regional Health Agency New Aquitaine (Other Government); University Hospital, Limoges (Other)
Responsible Party: Principal Investigator, Stephane Mandigout, Professor, Limoges University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SMandigout_ADEPINA
Record Dates: First submitted 2024-07-13; First posted 2024-08-16 (Actual); Last update posted 2024-08-16 (Actual); Status verified 2024-08

CONDITIONS: Chronic Disease; Chronic Condition; Stroke Sequelae; Age Problem; Parkinson Disease
Keywords: Physical training; Telerehabilitation; Fitness test; health professional; chronic disease
MeSH Terms: conditions — Chronic Disease; Parkinson Disease

STUDY DESIGN:
Intervention Model Description: Prospective pilot study.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Chronic disease patients (Experimental): The only intervention group (chronic disease patients) will use the ADEPINA device as part of their conventional treatment.
  Interventions: Device: Telerehabilitation intervention

INTERVENTIONS:
Device: Telerehabilitation intervention — Inclusion will take place within the framework of routine care for individuals with chronic diseases in rehabilitation services, hospitals, institutions, etc. The study will be offered to patients with chronic illnesses who are being cared for by their therapists. Data collection will be conducted in two sessions. The period between the two sessions will be determined based on the patient's availability, not exceeding a period of 12 weeks:
  1. 1st session at 0 week : Conducting activities and initial evaluation at their usual care center. Therapists will perform the various planned tests and evaluations.
  2. 2nd session at 12 weeks : This session will take place under the same conditions as the first one and without any potential health risks to the participants.
  3. A final evaluation will be carried out at the 18-week follow-up. A telephone call will be made between sessions to check in and assist participants in case of any issues during the study.

SUMMARY:
Exercise Rehabilitation (ER) is widely used and effective in the treatment of chronic diseases; however, patients do not adhere to ER programs. Tele-rehabilitation is effective and often used to support and improve patient adherence. Thus, the ADEPINA device could be a promising solution for the individualized management of patients by their therapists. The aim of the study will be: a) To assess functional improvement, measured by the 6-minute walk test (6MWT) after the 12 weeks ER program in people with chronic disease. Additionally, the study will assess the individualized program' adherence and his effect on patients' physical fitness and quality of life. Methods: Fifty patients will follow individualized ER sessions to their patients (with chronic diseases) using the ADEPINA device, 2 to 3 times per week for 12 weeks. At the end of the intervention, the investigator will assess patients' lower limb strength (with sit to stand test), dynamic balance (Timed up and go test), patients' adherence to the ER program by evaluating the usage time of the system by participants, the treatment credibility and participant expectations for improvement will be assessed with the French version of the Credibility and Expectancy Questionnaire. The investigator will also evaluate the patients' quality of life (using the "World Health Organization Quality of Life" (WHOQOL) scale) at the beginning and end of the intervention. Discussion: This interventional pilot study could have positive impacts for participants and explore gaps in the current literature regarding the individualized telerehabilitation program' feasibility.

DETAILED DESCRIPTION:
The ADEPINA project is a 12- week prospective multicentric pilot study. The project will be conducted by the HAVAE laboratory and the Limoges university will be the promoter. The study protocol is in accordance with the Standard Protocol Items Recommendations for Interventional Trials (SPIRIT) guidelines. Patients will perform ER program proposed by their professionals (as part of their routine care) through ADEPINA web platform for 12 weeks with evaluations before and after the intervention.

Participants recruitment:

The principal investigator will recruit ER therapists working in the private sector, public sector, or both. The investigator will present the study to potential participants. This study will be conducted with ER professionals (physiotherapists, kinesiologists) and their patients with chronic conditions. Volunteers who meet the inclusion criteria below and provide written consent will be included and will then receive an information notice.

Inclusion will take place within the framework of routine care for individuals with chronic diseases in rehabilitation services, hospitals, institutions, etc. The study will be offered to patients with chronic conditions who are being cared for by their therapists. Data collection will be conducted in two sessions. The period between the two sessions will be determined based on the patient's availability, not exceeding a period of 12 weeks:

1. 1st session at Day 0: Conducting activities and initial evaluation at their usual care center. Therapists will perform the various planned tests and evaluations.
2. 2nd session at 12 weks: This session will take place under the same conditions as the first one and without any potential health risks to the participants.
3. A final follow up session will be carried out at 18 weeks. A telephone call will be made between the two sessions to check in and assist participants (both therapists and patients with chronic illnesses) in case of any issues during the study. Recruitment will be coordinated by the clinical investigation center of the University Hospital of Limoges.

Eligibility:

Participants must meet the following criteria before being included in the present study. Professionals must: a) Be a physiotherapist or kinesiologist working in the public sector, private sector, or in a mixed capacity, b) Have been graduated for at least one year, c) Conduct RE with their patients and provide written consent.

The patients of the professionals included in the study must: a) Be 18 years of age or older, b) Be capable of giving informed consent, c) Be registered with the French social security system, e) Be under the care of a rehabilitation exercise professional.

Non inclusion criteria We will not include patients who: a) Have an intolerance or inability to use digital tools, b) Have a cognitive impairment, c) Have contraindications to physical activity (unstable diabetes, unstable hypertension, unstable angina, intracardiac thrombus). In addition, we will not include professionals who refuse to participate in the study.

Exclusion Criteria Participants will be excluded from the study if: a) They (patients or professionals) withdraw their consent to participate in this study during or after data collection, b) A serious adverse event occurs to a patient being treated by a professional included in the study (deterioration of the participant's health, fall, injury). All participants who request to leave the study will be excluded. Similarly, participants who do not use the platform before the final evaluation after two reminders will be excluded from this study and the final analysis.

Sample size calculation :

The sample size calculation is based on a previous study by Hwang et al., that assessed efficacy and safety of a group-based heart failure rehabilitation program delivered into each participant's home via an online telerehabilitation system. Investigators hypothesized that the 12 weeks telerehabilitation program would improve the attendance rates among patients after the intervention by 10%. In addition, a personalized telerehabilitation program could improve clinical parameters such as physical conditions (Timed up and go, sit to stand tests …) and quality of life. Investigators performed an estimation with 0.80 power and 0.05 α risk. The sample size required was 35 patients. Investigators added 20% to ensure the statistical power of the study, considering possible drop-out. The total sample will consist in 50 patients.

Ethical approval and considerations:

All procedures will follow the recommendations of the Good Clinical Practice Guidelines of the Declaration of Helsinki. This project will receive authorization from the ethics and individual protection committee (IFC) sud-est 2. Every significant amendment to the protocol will have to be approved by the Committee prior to its implementation. The study will also follow the principles of the Declaration of Helsinki. The results of the current study will be published in relevant scientific journals and be disseminated in international conferences. The consent form and the information notice will be drawn up in triplicate, one copy of which will be given to each participant. This study is part of routine care, and people with chronic diseases will be cared for in accordance with their usual care plan. Finally, the risks associated with this study are very low, because considering the "jardé law" in effect in France, this is interventional research on the human person with minor risk (RIPH3).

Intervention

ADEPINA device :

i. Web-based Platform Therapists will create physical training sessions by compiling exercises into video capsules for the patients. Patients will find these sessions in their personal spaces and will perform the same movements requested by the therapist, adhering to safety instructions and the prescribed dosage (repetitions, sets, etc.). Therapists will use equipment regularly utilized in routine care.

ii. Android Tablet All patients will have access to a tablet that allows them to view the sessions from their respective caregivers. They can also perform physical fitness tests by following the therapist's instructions.

iii. Wearable Sensor The evaluation of physical activity levels is conducted using tools from the wearable sensor, which includes MEMS components commonly found in smartwatches and mobile phones (accelerometer, gyrometer, magnetometer). Participants will need to wear the sensor on their wrist during evaluations (Sit to stand, TUG, etc.).

Training program We conceptualized our telerehabilitation device based on our previous studies regarding the acceptability of the ADEPINA device. According to previous studies, patients prefer their care to be provided by their healthcare professionals. Therefore, rehabilitation exercise professionals have the opportunity to design their own personalized rehabilitation exercise sessions for their patients. These professionals are required to adhere to the World Health Organization (WHO) recommendations regarding the design of rehabilitation exercise sessions.

Outcomes and Evaluations:

Primary outcomes Over a 12-weeks period, participants will use the digital platform for their regular rehabilitation exercise sessions. This will be a pilot study based on the collection and analysis of quantitative data. The study will investigate the functional improvement, measured by the 6-minute walk test (6MWT) after the 12 weeks ER program in people with chronic disease.

Secondary outcomes

In addition, the study will assess:

* The adherence to the rehabilitation exercise program will be assessed by evaluating the system usage time by participants (professionals and their patients). Specifically, we will examine program adherence through the rate of professionals and patients who completed the intervention and both evaluations at Day 0, Week 12 and Week 18.
* Lower limb muscles strength using the Sit-to-Stand Test (STS). Participants will be instructed to stand up completely and then sit down on a chair with their back against the backrest as quickly as possible within 30 seconds, while keeping their arms crossed over their chest. The number of repetitions performed during the 30-second STS test will be simultaneously recorded by our custom sensor, which was validated in our recent study. Performance on the STS test is associated with disability, fall risk, hip fractures, and mortality among elderly individuals and those with chronic diseases
* Quality of life will be assessed using the World Health Organization Quality of Life (WHOQOL) questionnaire.
* Patients' dynamic balance using the Timed Up and Go (TUG) test assesses functional mobility and dynamic balance in individuals. The subject rises from a chair, walks a distance of 3 meters, turns around, walks back, and sits down. Participants will be instructed to sit upright in the chair, hands on thighs, and back against the chair's backrest. Once the wearable sensor gives the starting signal, they will rise from the chair, walk at their normal pace, turn around just after passing the 3-meter mark, walk back, and sit down again. The test duration will be measured by our custom sensor, which was also validated in our recent study.
* The treatment credibility and participant expectations for improvement will be assessed with the French version of the Credibility and Expectancy Questionnaire (CEQ).

The CEQ includes a Credibility subscale (3 items) and an Expectancy subscale (3 items). The Credibility subscale has a 1-9 rating scale (1 "not at all" to 9 "very") for a total sub-score ranging from 3 to 27. The Expectancy scale has a 0-100% scale, and item 2 has a 1-9 rating scale for a total sub-score ranging from 3 to 27 after transforming the percentage scales. A moderate score ranges between 13.50 and 20.25; scores above 20.25 are considered high.

Statistical analysis:

Descriptive statistics, including frequencies, percentages, median and interquartile range, will be performed to examine the characteristics of the participants. For the qualitative part, a thematic analysis will be carried out to identify the salient aspects of health professionals' experiences and opinions regarding the ADEPINA device. At the end of the intervention, the average usability rate and the attractiveness of the platform to professionals and their patients will be assessed. We will compare clinical parameters before and after training (between Day 0 and week 12) using either the paired student's t test or the non-parametric Mann- Whitney test, depending on whether the data follow a normal distribution. Data will be analyzed with an analysis of variance (between Day 0, Week 12 and week 18).

All participants will be included in the analysis (intention-to-treat analysis). The quantitative analysis will be performed using SPSS V.23.0.0.3 (IBM® SPSS Statistics) and qualitative analysis will be performed by XLSTAT 16 software. The threshold of significance for all tests will be 0.05.

ELIGIBILITY:
Inclusion Criteria for professionals of exercise rehabilitation (ER):

* Be a physiotherapist or kinesiologist working in the public sector, private sector, or in a mixed capacity,
* Have been graduated for at least one year,
* Conduct ER program with chronic patients and provide written consent.

Inclusion Criteria for chronic patients :

* Be 18 years of age or older,
* Be able to walk with or without assistives devices
* Be capable of giving informed consent,
* Be registered with the French health social security system,
* Be under the care of a rehabilitation exercise professional.

Non-inclusion criteria for patients :

* Have an intolerance or inability to use digital tools,
* Have a cognitive impairment,
* Have contraindications to physical activity (unstable diabetes, unstable hypertension, unstable angina, intracardiac thrombus).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-01 (Estimated); Primary Completion 2026-12 (Estimated); Study Completion 2027-07 (Estimated)

PRIMARY OUTCOMES:
To assess functional improvement, measured by the 6-minute walk test (6MWT) after the 12 weeks ER program in people with chronic disease. | Day 0, Week 12, Week 18
  The investigator will assess the 6-minutes walk distance change after the intervention

SECONDARY OUTCOMES:
To evaluate the impact of the intervention on patient's lower limb strengh | Day 0, Week 12, Week 18
  Physical fitness will be assessed using a clinical test (a 30 seconde' sit to stand test) validated and standardized among the chronic disease population.
To evaluate the impact of the intervention on patient's dynamic balance | Day 0, Week 12, Week 18
  Physical fitness will be assessed using a clinical test (a time up and go test) validated and standardized among the chronic disease population.
To assess the impact of the intervention onpatient's quality of life | Day 0, Week 12, Week 18
  Quality of life will be assessed using the World Health Organization Quality of Life (WHOQOL) questionnaire
The adherence to the rehabilitation exercise program will be assessed by evaluating the system usage time by participants | Week 12, Week 18.
  Specifically, this study will examine program adherence through the rate of patients who completed the intervention sessions and evaluations
The treatment credibility and participant expectations for improvement were assessed with the French version of the Credibility and Expectancy Questionnaire (CEQ). | Week 12, Week 18.
  The CEQ includes a Credibility subscale (3 items) and an Expectancy subscale (3 items). The Credibility subscale has a 1-9 rating scale (1 "not at all" to 9 "very") for a total sub-score ranging from 3 to 27. The Expectancy scale has a 0-100% scale, and item 2 has a 1-9 rating scale for a total sub-score ranging from 3 to 27 after transforming the percentage scales. A moderate score ranges between 13.50 and 20.25; scores above 20.25 are considered high.

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hwang R, Bruning J, Morris NR, Mandrusiak A, Russell T. Home-based telerehabilitation is not inferior to a centre-based program in patients with chronic heart failure: a randomised trial. J Physiother. 2017 Apr;63(2):101-107. doi: 10.1016/j.jphys.2017.02.017. Epub 2017 Mar 14. PMID 28336297
- [Background] Batalik L, Dosbaba F, Hartman M, Konecny V, Batalikova K, Spinar J. Long-term exercise effects after cardiac telerehabilitation in patients with coronary artery disease: 1-year follow-up results of the randomized study. Eur J Phys Rehabil Med. 2021 Oct;57(5):807-814. doi: 10.23736/S1973-9087.21.06653-3. Epub 2021 Feb 23. PMID 33619944
- [Background] Wu YQ, Long Y, Peng WJ, Gong C, Liu YQ, Peng XM, Zhong YB, Luo Y, Wang MY. The Efficacy and Safety of Telerehabilitation for Fibromyalgia: Systematic Review and Meta-analysis of Randomized Controlled Trials. J Med Internet Res. 2023 Apr 25;25:e42090. doi: 10.2196/42090. PMID 37097721
- [Result] Scott Kruse C, Karem P, Shifflett K, Vegi L, Ravi K, Brooks M. Evaluating barriers to adopting telemedicine worldwide: A systematic review. J Telemed Telecare. 2018 Jan;24(1):4-12. doi: 10.1177/1357633X16674087. Epub 2016 Oct 16. PMID 29320966
- [Result] Mura A, Maier M, Ballester BR, De la Torre Costa J, Lopez-Luque J, Gelineau A, Mandigout S, Ghatan PH, Fiorillo R, Antenucci F, Coolen T, Chivite I, Callen A, Landais H, Gomez OI, Melero C, Brandi S, Domenech M, Daviet JC, Zucca R, Verschure PFMJ. Bringing rehabilitation home with an e-health platform to treat stroke patients: study protocol of a randomized clinical trial (RGS@home). Trials. 2022 Jun 20;23(1):518. doi: 10.1186/s13063-022-06444-0. PMID 35725616
- [Result] Seinsche J, de Bruin ED, Saibene E, Rizzo F, Carpinella I, Ferrarin M, Ifanger S, Moza S, Giannouli E. Feasibility and Effectiveness of a Personalized Home-Based Motor-Cognitive Training Program in Community-Dwelling Older Adults: Protocol for a Pragmatic Pilot Randomized Controlled Trial. JMIR Res Protoc. 2023 Nov 9;12:e49377. doi: 10.2196/49377. PMID 37943591
- [Result] Bohannon RW, Crouch R. Minimal clinically important difference for change in 6-minute walk test distance of adults with pathology: a systematic review. J Eval Clin Pract. 2017 Apr;23(2):377-381. doi: 10.1111/jep.12629. Epub 2016 Sep 4. PMID 27592691
- See also: Related Info — http://pubmed.ncbi.nlm.nih.gov/29320966/